CLINICAL TRIAL: NCT01855113
Title: COMPARISON OF THE PERCEPTION OF PAIN BETWEEN ORTHODONTIC TREATMENT WITH Invisalign ® AND TREATMENT WITH BRACKETS
Status: Completed | Type: Observational
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Hicham El-Khatib, Associate professor, Doctor of Dental Medecine, Université de Montréal
Other Study IDs: 13-031-CERES-D
Record Dates: First submitted 2013-03-13; First posted 2013-05-16 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: PAIN
Keywords: PAIN; ORTHODONTIC TREATMENT; INVISALIGN
MeSH Terms: conditions — Pain | interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- INVISALIGN®: those with an Invisalign® Treatment for orthodontic correction
  Interventions: Device: Invisalign
- braces: those with braces for orthodontic correction.

INTERVENTIONS:
Device: Invisalign
  Groups: INVISALIGN®

SUMMARY:
This study aims to compare the pain experienced by patients undergoing orthodontic treatment with Invisalign ® corrective aligners with that of patients undergoing orthodontic treatment with conventional braces. Because the aligners are removable, nearly invisible and don't involve metal that can irritate teeth and gums, we are expecting less pain in the Invisalign Treatment and less affectation of the quality of life.

DETAILED DESCRIPTION:
The aims of the study are to determine:

the presence of pain, the magnitude of pain, the duration of pain, and the location of pain.

The hypotheses of this study are:

* Treatment with Invisalign ® aligners result in less pain than the braces
* Treatment with Invisalign ® aligners result in less irritation to the soft tissues with braces
* Pain should increase each time the aligners are put in the mouse and decrease until disappearing on the third day.
* The quality of life will be most affected by treatment with braces than with Invisalign ®.
* Null Hypothesis: There is no difference at all points between the two treatments.

ELIGIBILITY:
Inclusion Criteria:

* In permanent dentition;
* Age less than 30 years;
* No medical contraindications or presence of systemic diseases (including nervous system disorders);
* No missing teeth except the third molars;
* Orthodontic treatment without extraction.
* Relationship skeletal cl. I (or slightly cl. II or cl. III)
* Speak and understand French without help.

Exclusion Criteria: lack of compliance with appointments.

-

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients are recruited from the Department of Orthodontics at the University of Montreal.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
PAIN DURING INVISALIGN TREATMENT | 6 MONTHS
  A questionnaire will be completed by the patient at different time points during treatment.
  This questionnaire includes questions on descriptive pain: location, duration, alteration in quality of life and a visual analog scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Hicham EL-Khatib, DMD,MSc, Study Director — Université de Montreal
Locations (1):
- clinique d'orthodontie de l'Université de Montréal, Montreal, Quebec, Canada